CLINICAL TRIAL: NCT00383903
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study of Safety, Reactogenicity and Immunogenicity of 2 or 3 Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus Vaccine at 10E6.5 CCID50 Viral Concentration in Healthy Infants (Approximately 5-10 Weeks Old) in the Republic of South Africa
Brief Title: Evaluate Safety & Immunogenicity of 2 or 3 Doses of GSK HRV Vaccine in Healthy Infants in South Africa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 444563/013
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Rotavirus
MeSH Terms: conditions — Rotavirus Infections

INTERVENTIONS:
Biological: HRV vaccine — Two or three oral doses

SUMMARY:
The purpose of this study is to determine the appropriate regimen of GSK HRV vaccine for concomitant administration with EPI vaccines to infants in South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants born after a normal gestation period (>=36 weeks), between 5 and 10 weeks of age at Dose 1 with confirmed negative HIV status of the subject's mother.
* Written informed consent was obtained from the parent/guardian of the subject before study entry.

Exclusion Criteria:

* History of allergic disease/polio disease,
* Confirmed or suspected immunosuppressive or immunodeficient condition,
* Clinically significant history of chronic gastrointestinal disease or other serious medical condition as determined by the investigator,
* Received treatment prohibited by the protocol.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.

Ages: 5 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 472 (Actual)
Dates: Start 2003-09; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Seroconversion after HRV vaccination

SECONDARY OUTCOMES:
shedding, serum anti-rota IgA antibody concentrations, anti-polio 1, 2 and 3 seroprotection rates, reactogenicity, safety

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- South Africa (6):
  - GSK Investigational Site, Brits
  - GSK Investigational Site, Ga-Rankuwa
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Pretoria North
  - GSK Investigational Site, Rooihuiskraal
  - GSK Investigational Site, Sunnyside, Pretoria

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Steele AD et al. Comparison of 2 different regimens (two doses versus three doses) in terms of reactogenicity and immunogenicity of the live attenuated human rotavirus vaccine Rotarix™ (RIX4414) in South African infants. Abstract presented at the 9th dsRNA Virus Meeting. Cape Town, South Africa, 21-26 Oct 2006.
- [Background] Steele AD et al. Comparison of 2 different regimens (two doses versus three doses) in terms of reactogenicity and immunogenicity of the live attenuated human rotavirus vaccine Rotarix™ (RIX4414) in South African infants. Abstract presented at ASCOOD. Bangkok, Thailand, 8-10 March 2006.
- [Background] Steele AD et al. Difference in immune responses between 2 different regimens of RIX4414 ( 106.5 CCID50 viral concentration) in South Africa. Abstract presented at the 4th World Congress of the World Society for Pediatric Infectious Diseases (WSPID). Warsaw, Poland, 01-04 Sept 2005.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 444563/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 444563/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 444563/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 444563/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 444563/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 444563/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register